CLINICAL TRIAL: NCT04815603
Title: A Phase 2a, 12-Week, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate Efficacy and Safety of BGE-117 in the Treatment of Anemia of Aging
Brief Title: Study to Evaluate Efficacy and Safety of BGE-117 in the Treatment of Anemia of Aging
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The program priority for execution of this clinical trial changed prior to enrollment of the first patient. The study was not withdrawn due to any safety concerns.
Sponsor: BioAge Labs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BGE-117-201
Record Dates: First submitted 2021-03-08; First posted 2021-03-25 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Anemia
Keywords: Anemia; BGE-117; BioAge
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- BGE-117 (Experimental): BGE-117 Capsules (4mg or 12mg) to be taken by mouth once a day for 84 days.
  Interventions: Drug: BGE-117
- Placebo (Placebo Comparator): Placebo Capsules to be taken by mouth once a day for 84 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BGE-117 — Active Treatment
  Arms: BGE-117
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The primary objectives of this study to evaluate the safety, tolerability and efficacy of BGE-117 in the treatment of anemia of aging in participants ≥ 65 years of age.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, multicenter, double- blind study of BGE-117 administered PO in participants ≥ 65 years of age for the treatment of anemia of aging. Anemia of aging accounts for approximately one-third of anemia in patients over 65 years of age, defined as a suboptimal hemoglobin level due to different underlying characteristics. This study's planned size is 160 evaluable subjects (80 subjects randomized to BGE-117 and 80 subjects randomized to placebo).

After signing informed consent, participants may be Pre-screened for hemoglobin using HemoCue, and subsequently will be screened for study eligibility. Screening will include full physical examination, vital signs, safety and study-related laboratory evaluation, ophthalmic exam, ECG, Wells score for DVT, and clinical outcome assessment. If confirmed that the participant qualifies for this protocol according to listed inclusion and exclusion criteria, participants will be randomized to BGE-117 or placebo, PO, once per day, for a treatment period duration of approximately 12 weeks. Dose adjustments for study medication during the treatment period are made according to a dosing algorithm to achieve and maintain hemoglobin (Hb) within the target range (12.5-13.0 g/dL). Study procedures and assessments are performed at various timepoints during the treatment period per the schedule outlined in the study protocol. Participants will undergo follow-up assessments for approximately 4 weeks after administration of the last dose.

ELIGIBILITY:
Inclusion Criteria:

* Ability to voluntarily provide written, signed, and dated informed consent to participate in the study
* An understanding, ability, and willingness to fully comply with study procedures and restrictions
* Is 65 years of age or older at the time of Screening (Visit 1)
* Anemia of Aging defined as a hemoglobin level in the range of ≥ 9.0 g/dL to ≤ 11.5 g/dL (≥ 90 g/L to ≤ 115 g/L) as determined by central laboratory measurement. (Note: For subjects with newly diagnosed anemia, appropriate investigations for the cause of the anemia should be completed according to standard-of-care under the direction of the subject's primary care physician.
* Weight at Screening (Visit 1) is ≥ 40.0 kg

Exclusion Criteria:

* History or diagnosis of any of the following:

  * Anemia due to pernicious anemia, thalassemia, sickle cell anemia, sickle trait, or myelodysplastic syndromes
  * Bone-marrow hypoplasia or pure red cell aplasia
  * Androgen deprivation therapy within the previous12 months or radiation treatment for prostate cancer
  * Thyroid-stimulating hormone (TSH) <0.1 mIU/L or >10.0 mIU/L
  * Folic acid and Vitamin B12 levels less than the lower limit of normal range
  * eGFR as measured by Modification of Diet in Renal Disease (MDRD) <30.0 mL/m/1.73 m2
  * Myocardial infarction, acute coronary syndrome, stroke, transient ischemic attack, or pro thrombotic arrhythmia or condition (e.g., untreated atrial fibrillation) within 6 months before Screening or during the Screening (Visit 1).
  * Cancer diagnosis with active or uncertain disease (i.e. active malignancy), or are receiving active treatment within 12 weeks before Screening (Visit 1) (squamous cell or basal cell carcinoma of the skin are excluded from this criterion)
  * Suspected or history of hematologic malignancy. Remote or childhood hematologic malignancies may be permitted as judged by the investigator. Age-related clonal changes in hematopoiesis (e.g., clonal hematopoiesis of indeterminate potential (CHIP), clonal cytopenia of undetermined significance (CCUS)) are permitted as judged by the investigator.
  * Intravenous (IV) iron within 12 weeks before Screening (Visit 1) or during the Screening Period or Treatment Period. Rescue therapy with IV iron is permitted during the Follow-up Period if the subject's hemoglobin is below their baseline level. Note: oral iron supplementation is permitted. The subject must have started treatment with oral iron supplements at least 4 weeks before Screening. The same dose and dosing regimen should be maintained throughout the Screening Period and Treatment Period.
* Erythropoieisis-stimulating agent (ESA) treatment within 12 weeks before Screening (Visit 1) or during the Screening Period or Treatment Period. Rescue therapy with ESA is permitted during the Follow-up Period if the subject's hemoglobin level is below baseline.
* History of uncontrolled hypertension including:

  * Difficult-to-control hypertension (unless approved by the investigator and the Medical Monitor)
  * Malignant hypertension (unless approved by the investigator and the Medical Monitor)
  * Systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 95 mmHg (confirmed by repeated measurement) within 2 weeks before randomization. Note:

    * Subjects being treated for hypertension should have been on a stable medication and dosing regimen for at least 8 weeks before randomization
    * Subjects may be rescreened after their blood pressure is controlled
* Evidence of gastrointestinal bleeding within 12 weeks before Screening (Visit 1), as judged by the investigator
* Blood or plasma donation within 8 weeks before Screening (Visit 1) or at any time during the study period.
* Class III heart failure, as defined by the New York Heart Association (NYHA) functional classification system
* QTcF > 500 msec or QTcF > 530 msec in subjects with bundle branch block Note: This evaluation will be done only at Screening (Visit 1); ECG and corresponding intervals and overall interpretation can be mechanically or manually read by an appropriately designated and trained personnel.
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≥ 3 × the upper limit of normal (ULN)
* Bilirubin > 1.5 × ULN (isolated bilirubin > 1.5 × ULN is acceptable if bilirubin is fractionated and direct bilirubin is < 35%) Note: Bilirubin increases associated with Gilbert's syndrome are permitted.
* A reported average intake of alcohol of ≥ 80 g/day (i.e., equivalent of 6 cans of beer or 5 shots of hard liquor)
* Increase in hemoglobin level to the target range (12.5-13.0 g/dL) would pose an unacceptable medical risk to the subject, as judged by the investigator
* History of severe allergic or anaphylactic reactions or hypersensitivity to excipients in the investigational product
* Use of another investigational agent within 30 days or 5 half-lives of the investigational agent; whichever is longer
* Prior randomization in the current study (BGE-117-201)
* Any current unstable medical condition that the investigator considers would put the subject at unacceptable risk, affect study compliance, or prevent the understanding of the study's objectives or investigational procedures or possible consequences. This includes:

  * Current, unstable active liver or biliary disease (generally defined by the onset of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal/gastric varices, persistent jaundice, or cirrhosis) Note: Stable liver disease (including asymptomatic gallstones, asymptomatic chronic hepatitis B, chronic hepatitis C, or Gilbert's syndrome) is acceptable if the subject otherwise meets entry criteria and the investigator and Sponsor approve entry into the study.
  * Current or relevant history of a medical condition that may require inpatient treatment or make the subject unlikely to complete the study
* Unable or unwilling to adhere to the contraception requirements specified in the protocol

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin | Day 85
  Change in Hemoglobin compared to baseline

SECONDARY OUTCOMES:
Functional Assessment of Chronic Illness Therapy-Fatigue Scale (FACIT-Fatigue) Score | Day 29, 57, 85 and Follow-up (up to 120 days)
  Improvement in FACIT-Fatigue Score compared to baseline. The FACIT-Fatigue assessment is a 13-item questionnaire that assesses self-reported fatigue and its impact on daily activities and function. The scale is scored from 0 (Not at all) to 4 (Very Much). A lower score is considered improvement and a better outcome.
Hemoglobin | Day 29, 57, and Follow-up (up to 120 days)
  Change in Hemoglobin compared to baseline
Short Physical Performance Battery (SPPB) Score | Day 29, 57, 85, and Follow-up (up to 120 days)
  Change in SPPB Score compared to baseline. The SPPB assessment consists of a Balance Test, a Gait Speed Test, and a Chair Stand Test. Each of the three tests is scored from 0 to 4 points with a composite score from 0 to 12 points. A higher score is considered a better outcome.
6-minute Walk Test (6MWT) Distance | Day 29, 57, 85, and Follow-up (up to 120 days)
  Change in 6MWT Distance compared to baseline. Increased distance is considered a better outcome.
36-Item Short Form Survey Instrument (SF-36) | Day 29, 57, 85, and Follow-up (Up to 120 days)
  Change in SF-36 compared to baseline. The SF-36 is a general health status questionnaire to assess patient perception of health in several domains, including physical functioning, role physical, bodily pain, vitality, social functioning, role emotional, mental health, and general health over the past 7 days. Each of the categories is scored from 0 to 100. A higher score is considered a better outcome.
BGE-117 Starting Dose Evaluation | First dose to Day 85
  Evaluate the starting dose of BGE-117 in the treatment of anemia of aging for subjects with eGFR ≥ 60 mL/min/1.73 m2 and subjects with eGFR ≥ 30 and < 60 mL/min/ 1.73 m2
Grip Strength | Day 29, 57, 85, and Follow-up (Up to 120 days)
  Evaluate the change in grip strength measures using the Jamar Hand Dynamometer grip strength test.
Clinical Global Impression (CGI) Measures | Day 29, 57, 85, and Follow-up (Up to 120 days)
  Change in CGI measures compared to baseline. The CGI is a questionnaire-based instrument to assess subjects' progress and treatment response over time. The study will collect the CGI-Change of Condition to measure change in energy level and CGI-Therapeutic Efficacy to assess perceived therapeutic efficacy of treatment. A lower score is considered a better outcome.

OTHER OUTCOMES:
Analysis of Pharmacokinetic Parameters to Develop a Population Pharmacokinetic Model for BGE-117 (AUC(0-24)/dose) | Day 1, 29, 57, and 85
  Single blood samples for pharmacokinetic analysis will be collected just prior to first dose and on Days 29, 57 and 85. Time of last dose and time of blood draw will be collected and these data will be used to attempt to develop a population pharmacokinetic model of BGE-117. If possible, AUC(0-24)/dose will be determined. Age, gender and renal function will be explored as covariates.
Analysis of Pharmacokinetic Parameters to Develop a Population Pharmacokinetic Model for BGE-117 (Clearance) | Day 1, 29, 57, and 85
  Single blood samples for pharmacokinetic analysis will be collected just prior to first dose and on Days 29, 57 and 85. Time of last dose and time of blood draw will be collected and these data will be used to attempt to develop a population pharmacokinetic model of BGE-117. If possible, clearance will be determined. Age, gender and renal function will be explored as covariates.
Analysis of Pharmacokinetic Parameters to Develop a Population Pharmacokinetic Model for BGE-117 (Volume of Distribution) | Day 1, 29, 57, and 85
  Single blood samples for pharmacokinetic analysis will be collected just prior to first dose and on Days 29, 57 and 85. Time of last dose and time of blood draw will be collected and these data will be used to attempt to develop a population pharmacokinetic model of BGE-117. If possible, volume of distribution will be determined. Age, gender and renal function will be explored as covariates.
Analysis of Pharmacokinetic Parameters to Develop a Population Pharmacokinetic Model for BGE-117 (Half-Life) | Day 1, 29, 57, and 85
  Single blood samples for pharmacokinetic analysis will be collected just prior to first dose and on Days 29, 57 and 85. Time of last dose and time of blood draw will be collected and these data will be used to attempt to develop a population pharmacokinetic model of BGE-117. If possible, half-life will be determined. Age, gender and renal function will be explored as covariates.
Safety Analyses (Treatment-Emergent Adverse Events) - Number of Events | First Dose to Day 85 and Follow-up (Up to 120 days)
  Safety analyses will be performed based on the corresponding Safety Set. The number of events of treatment-emergent AEs (TEAEs) will be calculated overall by system organ class, preferred term, and treatment group for each cohort and treatment group. The number of subjects with TEAEs will be further summarized by severity and relationship to the IP.
Safety Analyses (Treatment-Emergent Adverse Events) - Incidence | First Dose to Day 85 and Follow-up (Up to 120 days)
  Safety analyses will be performed based on the corresponding Safety Set. The incidence of treatment-emergent AEs (TEAEs) will be calculated overall by system organ class, preferred term, and treatment group for each cohort and treatment group. The number and percentage of subjects with TEAEs will be further summarized by severity and relationship to the IP.
Safety Analyses (Treatment-Emergent Adverse Events) - Percentage | First Dose to Day 85 and Follow-up (Up to 120 days)
  Safety analyses will be performed based on the corresponding Safety Set. The percentage of treatment-emergent AEs (TEAEs) will be calculated overall by system organ class, preferred term, and treatment group for each cohort and treatment group. The percentage of subjects with TEAEs will be further summarized by severity and relationship to the IP.
Safety Analyses (Adverse Events) - Individual Summary | First Dose to Day 85 and Follow-up (Up to 120 days)
  Adverse events related to IP, AEs leading to withdrawal, SAEs, and deaths will be summarized/listed as part of the overall analysis of safety.
Safety Analyses (Quantitative Safety Data) - Clinical Laboratory Tests | First Dose to Day 85 and Follow-up (Up to 120 days)
  Clinical laboratory tests (Complete Blood Count, Serum Clinical Chemistries, Coagulation and D-Dimer, Erythropoietin, Hemoglobin Electrophoresis, Inflammation Panel, Iron Panel, Folate and Vitamin B12, Lipid Panel, Thyroid, Urinalysis, Fecal Occult Blood Test) findings will be summarized by treatment group and visit. Descriptive statistics will be calculated for quantitative safety data as well as for the difference from baseline, if applicable. Frequency counts will be compiled for the classification of qualitative safety data. The baseline for safety data will be defined as the last value prior to the first dose of IP. Potentially clinically important findings will also be summarized or listed.
Safety Analyses (Quantitative Safety Data) - Vital Signs | First Dose to Day 85 and Follow-up (Up to 120 days)
  Vital signs (systolic and diastolic blood pressure and pulse rate) findings will be summarized by treatment group and visit. Descriptive statistics will be calculated for quantitative safety data as well as for the difference from baseline, if applicable. Frequency counts will be compiled for the classification of qualitative safety data. The baseline for safety data will be defined as the last value prior to the first dose of IP. Potentially clinically important findings will also be summarized or listed.
Safety Analyses (Quantitative Safety Data) - Ophthalmology Examinations | First Dose to Day 85 and Follow-up (Up to 120 days)
  Ophthalmology examinations findings will be summarized by treatment group and visit. The assessment will include measurement of best-corrected visual acuity, intraocular pressure, anterior aqueous chamber examination, and fundoscopic examination. Descriptive statistics will be calculated for quantitative safety data as well as for the difference from baseline, if applicable. Frequency counts will be compiled for the classification of qualitative safety data. The baseline for safety data will be defined as the last value prior to the first dose of IP. Potentially clinically important findings will also be summarized or listed.
Safety Analyses (Quantitative Safety Data) - Wells Score for DVT | First Dose to Day 85 and Follow-up (Up to 120 days)
  The Well's Criteria will be used to evaluate for the presence of deep vein thrombosis (DVT) and summarized by treatment group and visit. Descriptive statistics will be calculated for quantitative safety data as well as for the difference from baseline, if applicable. Frequency counts will be compiled for the classification of qualitative safety data. The baseline for safety data will be defined as the last value prior to the first dose of IP. Potentially clinically important findings will also be summarized or listed.
Safety Analyses (Quantitative Safety Data) - Electrocardiogram (ECG) | First Dose to Day 85 and Follow-up (Up to 120 days)
  Electrocardiogram (ECG) will be performed with heart rate, PR, QRS, and QT (pre-corrected) intervals will be measured and QTcF will be calculated. ECG findings will be summarized by treatment group and visit. Descriptive statistics will be calculated for quantitative safety data as well as for the difference from baseline, if applicable. Frequency counts will be compiled for the classification of qualitative safety data. The baseline for safety data will be defined as the last value prior to the first dose of IP. Potentially clinically important findings will also be summarized or listed.
Correlation of HemoCue to Central Laboratory Hemoglobin Values | Pre-Screening to Day 78
  Compare the Hemoglobin values obtained using the HemoCue system to the Hemoglobin values obtained from blood samples tested by the central laboratory.

CONTACTS AND LOCATIONS:
Locations (13):
- Australia (13):
  - Paratus Clinical Research - Western Sydney, Blacktown, New South Wales
  - Emeritus Research Sydney, Botany, New South Wales
  - Northern Beaches Clinical Research, Brookvale, New South Wales
  - Vale Medical Practice, Brookvale, New South Wales
  - Paratus Clinical Research Central Coast, Kanwal, New South Wales
  - Browns Plains Family (Sonic/IPN), Browns Plains, Queensland
  - Parkwood Family Practice (Sonic/IPN), Gold Coast, Queensland
  - AusTrials Taringa, Taringa, Queensland
  - AusTrials Wellers Hill, Tarragindi, Queensland
  - PARC Clinical Research, Adelaide, South Australia
  - Casey Superclinic (Sonic/IPN), Berwick, Victoria
  - Emeritus Research - Camberwell, Camberwell, Victoria
  - Camberwell Road Medical Practice (Sonic/IPN), Hawthorn E., Victoria

IPD SHARING:
Plan to Share IPD: No